CLINICAL TRIAL: NCT02723045
Title: The Comparison of the Quality of Life and Outcomes in Patient's With Reducible Inguinal Hernias: Laparoscopic Totally Extra-peritoneal (TEP) Versus Modified Lichtenstein Hernioplasty
Brief Title: Quality of Life of TEP vs Lichtenstein Hernioplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sarawak General Hospital (Other)
Responsible Party: Principal Investigator, Siow Sze Li, General Surgeon, Sarawak General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMRR-16-277-29543
Record Dates: First submitted 2016-03-14; First posted 2016-03-30 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Inguinal Hernia
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open modified Lichtenstein repair (Active Comparator): Patients will undergo open repair of their inguinal hernias
  Interventions: Procedure: Open Lichtenstein Hernioplasty
- Laparoscopic TEP inguinal hernia repair (Active Comparator): Patients will undergo laparoscopic repair of their inguinal hernias
  Interventions: Procedure: Laparoscopic TEP Hernioplasty

INTERVENTIONS:
Procedure: Open Lichtenstein Hernioplasty
  Arms: Open modified Lichtenstein repair
Procedure: Laparoscopic TEP Hernioplasty
  Arms: Laparoscopic TEP inguinal hernia repair

SUMMARY:
To determine if there is a difference in the quality of life in between patients who undergoes laparoscopic totally extra-peritoneal (TEP) or modified Lichtenstein hernioplasty

DETAILED DESCRIPTION:
Patients presenting with reducible inguinal hernias will be randomized between open or laparoscopic repair groups. The primary outcome will be the quality of life scores. Patients will be followed-up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Both genders
* Unilateral inguinal hernias
* Reducible inguinal hernias
* Elective setting

Exclusion Criteria

* ASA Physical Status (American Society of Anaesthesiologists) Grade > 2
* Recurrence
* Inguinal-scrotal hernias
* Prostatectomy, Pfannenstiel incision, previous pre-peritoneal surgery
* Pregnancy
* Refusal for general anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-10 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Quality of life | 12 months
  Carolina Comfort Scale

SECONDARY OUTCOMES:
Operating time | 12 months
Duration of hospitalization | 12 months
Complications | 12 monthts
Recurrence | 12 months
  Recurrence of hernia after repair

IPD SHARING:
Plan to Share IPD: No